CLINICAL TRIAL: NCT05382039
Title: Effects of Electrotherapy on Cervical Spine Proprioception, Pain, Anxiety, and Disability in Adults With Subclinical Neck or Upper Quadrant Pain.
Brief Title: Effects of Electrotherapy on Pain, Anxiety, Motion and Disability in Adults With Neck or Upper Body Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Eric Johnson, Associate Director, Doctor of Physical Therapy Program & Director, Neuroscience Research Laboratory, Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5220149
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
Keywords: Neck, upper quadrant, upper body, chronic pain, sub-clinical pain, mild pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Subjects without Pain (No Intervention): This group will include twenty participants with no neck and/or upper quadrant pain that will not receive transcutaneous electrical nerve stimulation treatment.
- Subjects with Pain and No Intervention (No Intervention): This group will include twenty participants with neck and/or upper quadrant pain that will not receive transcutaneous electrical nerve stimulation treatment.
- Subjects with Pain and Intervention (Experimental): This group will include twenty participants with neck and/or upper quadrant pain that will receive transcutaneous electrical nerve stimulation treatment.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — High frequency sensory transcutaneous electrical nerve stimulation
  Arms: Subjects with Pain and Intervention

SUMMARY:
This will be a prospective randomized controlled trial with sixty adults, 20 to 40 years of age. There will be three groups as follows: the normal group, control group, and intervention group where subjects will receive instructions for home use of TENS for pain reduction. The aim is for an equal distribution of males and females in each group.

DETAILED DESCRIPTION:
This will be a prospective randomized controlled trial with sixty adults, 20 to 40 years of age. There will be three groups as follows: twenty subjects with no pain in the normal group; forty subjects with chronic subclinical neck or upper quadrant pain will be randomized into two groups: twenty subjects in the control group, and twenty subjects in the intervention group. The aim is for an equal distribution of males and females in each group.

Data will be collected for each subject using the NORAXON® myoMOTION™ System, the visual analog scale (VAS), the State-Trait Anxiety Inventory (STAI), and the Neck Disability Index (NDI); all assessments will be made by a clinician.

Normal group (20 subjects): Initial assessment on day one and post assessments on day eight and on day thirty. Control group (20 subjects): Initial assessment on day one and post assessments on day eight and on day thirty. Intervention group (20 subjects): Initial assessment on day one pre-intervention and post-intervention assessment of high-frequency sensory TENS (gate control theory of pain) for thirty minutes followed by post-assessments in day eight and day thirty.

The intervention group will receive a thirty-minute high frequency TENS (gate control theory of pain) once a day for seven days and twenty-one days after the initial seven days to measure immediate and short-term effects on the dependent variables further described below. Subjects will be educated on TENS usage by a licensed physical therapist. A daily log will be given to all subjects in the intervention group to assure compliance with treatment. In addition, the TENS device will keep track of date, time and day of usage, and TENS parameters.

ELIGIBILITY:
Inclusion Criteria for Subjects without Pain Group:

* > 19 and <41 years of age
* Currently enrolled as students at Loma Linda University.
* No pain

Exclusion Criteria for Control Group:

* Neck and/or upper quadrant pain
* <20 years or >40 years of age

Inclusion Criteria for Subjects with Pain Groups:

* >19 and <41 years of age
* Currently enrolled as students at Loma Linda University
* No acute pain
* With neck and/or upper quadrant chronic pain
* With <5/10 pain on the Visual Analog Scale (VAS)

Exclusion Criteria for Subjects with Pain Groups:

* <20 years or >40 years of age
* Acute pain
* With >5/10 pain on the Visual Analog Scale (VAS)
* Currently receiving clinical pain treatment
* Pain medications within six hours of data collection
* Contraindications for the use of electrotherapy

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Johnson, DSc, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Without Pain: This group included twenty participants with no neck and/or upper quadrant pain that did not receive transcutaneous electrical nerve stimulation treatment.
- Subjects With Pain and No Intervention: This group included twelve participants with neck and/or upper quadrant pain that did not receive transcutaneous electrical nerve stimulation treatment.
- Subjects With Pain and Intervention: This group included eleven participants with neck and/or upper quadrant pain that did receive transcutaneous electrical nerve stimulation treatment.
  Transcutaneous Electrical Nerve Stimulation: High frequency sensory transcutaneous electrical nerve stimulation
Period: Overall Study
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention
Started | 21 | 12 | 12
Completed | 16 | 12 | 10
Not Completed | 5 | 0 | 2
Not completed — Score on pain scale was not zero. Subjects randomized to this arm had to have zero pain. | 5 | 0 | 0
Not completed — One subject unable to return for reassessment as required by protocol timeline. | 0 | 0 | 1
Not completed — waiting for confirmation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Unable to analyze 7 subjects due to:
  * 1 subject (pain and intervention) unable to return after two weeks for reassessment.
  * 1 subject (pain and intervention) unable to complete data collection due to a pain score VAS >4/10.
  * 1 subject (no pain) unable to complete data due to lightheadedness.
  * 4 subjects (no pain) excluded due to a pain score >0/10.
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention | Total
Number analyzed (Participants) | 16 | 12 | 10 | 38
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 subject (pain and intervention) unable to return after two weeks for reassessment.
  1 subject (pain and intervention) unable to complete data collection due to a pain score VAS >4/10.
  1 subject (no pain) unable to complete data due to lightheadedness. 4 subjects (no pain) excluded due to a pain score >0/10.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 16 | 12 | 10 | 38
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Unable to analyze 7 subjects due to:
  1 subject (pain and intervention) unable to return after two weeks for reassessment.
  1 subject (pain and intervention) unable to complete data collection due to a pain score VAS >4/10.
  1 subject (no pain) unable to complete data due to lightheadedness. 4 subjects (no pain) excluded due to a pain score >0/10.
  Participants
    Female | 12 | 11 | 5 | 28
    Male | 4 | 1 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Chronic Subclinical Neck or Upper Quadrant Pain
Description: Assessed with the Visual Analog Scale (VAS) which is a subjective measure of pain intensity consisting of a 10 centimeter (cm) line with anchor statements on the left (no pain) and extreme pain on the right. Pain scores will be determined by measuring the distance in cm from "no pain" or 0 cm to the participant's anchor point.
Time Frame: Change between baseline and two weeks from time of enrollment
Population: 16 subjects (without pain) were analyzed that reflects outcome measure below
Measure: Median (Full Range); unit: cm
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention
Number analyzed (Participants) | 16 | 12 | 10
cm | 0 [0 to 0] | 2.0 [0.1 to 3.8] | 2.0 [0.1 to 3.8]

2. Secondary Outcome: Neck Proprioception
Description: Measurements assessed with NORAXON® myoMOTION™ System that is a composite measurement through an instrument that utilizes inertial measurement units (IMUs) to measure angles of motion in joints via sensors place on the head and neck. This system will measure cervical spine proprioception utilizing the joint position error (JPE) test by indicating the ability of a blindfolded subject to accurately reposition their head back to a predetermined neutral point after head movement.
Time Frame: Baseline
Population: 16 subjects (without pain) were analyzed that reflects outcome measure below
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention
Number analyzed (Participants) | 16 | 12 | 10
degrees | 4.2 (2.3) | 4.7 (4.2) | 4.7 (4.2)

3. Secondary Outcome: Level of Anxiety
Description: Assessed with the State-Trait Anxiety Inventory-form Y (STAI) which is a definitive clinical composite measure of state and trait anxiety in adults. Form Y has 20 items for assessing trait anxiety and 20 for state anxiety which will indicate how the subject feels "right now"/"at this moment" and how the subject "generally feels." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always") for a potential total of 80 points. A score of zero points represents no anxiety. A score of 80 points represents severe anxiety.
Time Frame: Change between baseline and two weeks post-enrollment
Population: 16 subjects (without pain) were analyzed that reflects outcome measure below
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention
Number analyzed (Participants) | 16 | 12 | 10
score on a scale | 13.5 (4.8) | 18.0 (7.0) | 18.0 (7.0)

ADVERSE EVENTS:
Time Frame: 2 weeks post enrollment
Description: No adverse events noted
Groups:
- Subjects Without Pain: This group included sixteen participants with no neck and/or upper quadrant pain that did not receive transcutaneous electrical nerve stimulation treatment.
- Subjects With Pain and Intervention: This group included ten participants with neck and/or upper quadrant pain that did receive transcutaneous electrical nerve stimulation treatment.
  Transcutaneous Electrical Nerve Stimulation: High frequency sensory transcutaneous electrical nerve stimulation
Arm/Group | Subjects Without Pain | Subjects With Pain and No Intervention | Subjects With Pain and Intervention
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT05382039/Prot_002.pdf
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT05382039/SAP_003.pdf